CLINICAL TRIAL: NCT02449915
Title: Does Liposomal Bupivacaine Improve Pain Following Robotic Sacrocolpopexy and Rectocele Repair for Pelvic Organ Prolapse? A Randomized Placebo Controlled Trial
Brief Title: Improvement of Pain Following Robotic Sacrocolpopexy and Rectocele Repair for Pelvic Organ Prolapse
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 14-079
Record Dates: First submitted 2015-05-18; First posted 2015-05-20 (Estimated); Results first posted 2017-12-08 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-11

CONDITIONS: Pelvic Organ Prolapse
Keywords: sacrocolpopexy; rectocele repair
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Bupivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bupivacaine Arm (Experimental): Those subjects in the liposomal bupivacaine arm will have 30mL dilutional volume injected. Ten mL will be injected into the perineum in the posterior vaginal area and 20 mL will be injected the port site wounds in the abdomen (5 sites, 4 ml per incision).
  Interventions: Drug: Bupivacaine
- Placebo Arm (Placebo Comparator): Those subjects in the placebo arm will have 30 mL sterile normal saline injected. Ten mL will be injected into the perineum in the posterior vaginal area and 20 mL will be injected into the port site wounds in the abdomen (5 sites, 4 mL per incision).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bupivacaine — At the completion of the procedure, and at least 20 minutes after the injection of lidocaine with epinephrine (routine for the surgical procedure), those subjects in the liposomal bupivacaine arm will have 30mL dilutional volume injected. Ten mL will be injected into the perineum in the posterior vaginal area and 20 mL will be injected the port site wounds in the abdomen (5 sites, 4 ml per incision).
  Other Names: Exparel
  Arms: Bupivacaine Arm
Drug: Placebo — At the completion of the procedure, and at least 20 minutes after the injection of lidocaine with epinephrine (routine for the surgical procedure), those subjects in the placebo arm will have 30mL total volume injected. Ten mL will be injected into the perineum in the posterior vaginal area and 20 mL will be injected the port site wounds in the abdomen (5 sites, 4 ml per incision).
  Other Names: Normal Saline
  Arms: Placebo Arm

SUMMARY:
To determine if the injection of liposomal bupivacaine to laparoscopic port sites and rectocele repair incisions at the completion of a robotic sacrocolpopexy with concomitant rectocele repair will result in decreased postoperative pain compared to injection of placebo.

DETAILED DESCRIPTION:
In the last 20 years, laparoscopic surgery has assumed an important role in gynecological surgery. Unfortunately, patient surveys indicate there has been little improvement in the incidence and severity of postsurgical pain in the past two decades. Postoperative pain is a common complaint, occurring in 5-15% of patients and has been shown to significantly contribute to overall patient dissatisfaction. It can lead to increased consumption of opioids, with subsequent nausea, delayed bowel function, and prolonged postoperative recovery. In an attempt to address pain related complications with port-site wounds, various methods of pain control have been attempted. Currently, no standard of care exists and management is based on surgeon and anesthesiologist preferences.

This study seeks to determine if the injection of liposomal bupivacaine to laparoscopic port sites and rectocele repair incisions at the completion of a robotic sacrocolpopexy with concomitant rectocele repair will result in decreased postoperative pain compared to injection of placebo.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older
* Planning for surgical treatment of POP with robotic sacrocolpopexy and rectocele repair under general anesthesia
* Patient undergoing concurrent hysterectomy and/or sub-urethral sling will be included

Exclusion Criteria:

* Pregnant or nursing
* Allergy to bupivacaine
* History of drug/alcohol abuse
* Severe cardiovascular, hepatic, renal disease, or neurological impairment
* Long-acting opioid use within 3 days or any opioid use within 24 hours before surgery
* Contraindication to: acetaminophen, oxycodone, non-steroidal anti- inflammatory drugs (NSAID)
* Administration of an investigational drug within 30 days before study
* Chronic pain syndromes
* Daily NSAID/opioid use
* Patients not undergoing general anesthesia
* Patients undergoing concurrent transvaginal mesh removal, anal sphincteroplasty, or fistula repair

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Pauls, MD, Principal Investigator — Cincinnati Urogynocolgy Associates
Locations (1):
- Cincinnati Urogynecology Associates, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Yeung J, Crisp CC, Mazloomdoost D, Kleeman SD, Pauls RN. Liposomal Bupivacaine During Robotic Colpopexy and Posterior Repair: A Randomized Controlled Trial. Obstet Gynecol. 2018 Jan;131(1):39-46. doi: 10.1097/AOG.0000000000002375. PMID 29215511

RESULTS

PARTICIPANT FLOW:
Groups:
- Bupivacaine Arm: Receiving 30mL dilutional volume of liposomal bupivacaine at the completion of the procedure, and at least 20 minutes after the injection of lidocaine with epinephrine (routine for the surgical procedure)
- Placebo Arm: Receiving 30 mL volume of sterile normal saline at the completion of the procedure, and at least 20 minutes after the injection of lidocaine with epinephrine (routine for the surgical procedure)
Period: Overall Study
Arm/Group | Bupivacaine Arm | Placebo Arm
Started | 35 | 35
Completed | 33 | 31
Not Completed | 2 | 4
Not completed — Exclusion criteria - drug use | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Intraoperative surgical findings | 1 | 1
Not completed — Abnormal preop lab | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Bupivacaine Arm: Receiving 30mL dilutional volume of the liposomal bupivacaine at the completion of the procedure, and at least 20 minutes after the injection of lidocaine with epinephrine (routine for the surgical procedure)
- Placebo Arm: Receiving 30 mL sterile normal saline at the completion of the procedure, and at least 20 minutes after the injection of lidocaine with epinephrine (routine for the surgical procedure)
- Total: Total of all reporting groups
Arm/Group | Bupivacaine Arm | Placebo Arm | Total
Number analyzed (Participants) | 33 | 31 | 64
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64 [57 to 68] | 61 [54 to 70] | 62 [55.3 to 68]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female only | 33 | 31 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 33 | 30 | 63
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 33 | 31 | 64

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scales (VAS) for Pain at 18 Hours Postoperatively
Description: VAS is a validated 100 millimeter scale with no pain as 0 mm and worst pain as 100 mm. Subjects drew a vertical line on the scale corresponding to their pain level.
Time Frame: 18 hours after surgery
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Bupivacaine Arm | Placebo Arm
Number analyzed (Participants) | 33 | 31
mm | 15.0 [1 to 35] | 20.5 [2.75 to 41.5]
Statistical Analysis 1: Comparison: Bupivacaine Arm vs Placebo Arm; Test type: Other; p = 0.52, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: From time of surgery to 12 weeks after surgery
Arm/Group | Bupivacaine Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/31
Other Adverse Events (participants affected / at risk) | 0/33 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes